CLINICAL TRIAL: NCT06468267
Title: Reduced Intensity Conditioning With Thiotepa Combined With Busulfan, Fludarabine and Cytarabine in Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Relapsed or Refractory Peripheral T-cell Lymphoma.
Brief Title: RIC With Thiotepa Combined With Bu/Flu/Ara-C in Allo-HSCT for Relapsed or Refractory PTCL.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xianmin Song, MD (Other)
Responsible Party: Sponsor-Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-202402-THI-FAB
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T cell lymphoma; reduced intensity conditioning regimen; thiotepa
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Thiotepa; fludarabine; Busulfan; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention arm (Experimental): Participants will receive allogenetic hematopoietic stem cell transplantation (allo-HSCT) with the reduced intensity conditioning regimen including thiotepa(5mg / kg / d-7d ( 1d )), fludarabine (30mg / m2 / d, -6d--2d ( 5d )), Ara-C (1g / m2 / d, -6d--2d ( 5d )), and busulfan(3.2mg / kg / d, -4d-3d ( 2d )).
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — The reduced intensity conditioning regimen is composed by thiotepa (5mg / kg / d-7d (1d)), fludarabine (30mg / m2 / d, -6d--2d (5d)), Ara-C (1g / m2 / d, -6d--2d (5d)), and busulfan (3.2mg / kg / d, -4d-3d (2d)).
  Other Names: fludarabine; busulfan; Cytarabine

SUMMARY:
This study is a single-center, single-arm, prospective phase II clinical trial that evaluates the efficacy and safety of an reduced-intensity conditioning (RIC) regimen with thiotepa combined with busulfan, fludarabine, and cytarabine for allogeneic hematopoietic stem cell transplantation in the treatment of relapse and refratory peripheral T-cells lymphoma. The conditioning regimen includes thiotepa at a dose of 5mg/kg/d at d -7 (1 day), fludarabine at 30mg/m2/d from d -6 to d -2 (5 days), cytarabine at 1g/m2/d from d -6 to d -2 (5 days), and busulfan at 3.2mg/kg/d from d -4 to d -3 (2 days). Conditioning begins on day -7, and donor hematopoietic stem cell infusion is performed on day 0. All patients will undergo bone marrow examination on day 14 and day 28 post-transplant, followed by bone marrow examinations every 30 days within the first year after transplantation, and every 60 days within the second year after transplantation. FDG-PET/CT imaging will be adopted every 6 months after transplantation. If disease relapse is suspected during the follow-up period, bone marrow and relapse site examinations will be conducted at any time. The primary study endpoints are the 1-year and 2-year progression-free survival (PFS) rates post-transplant. Secondary study endpoints include the incidence of acute graft-versus-host disease (GVHD) within 180 days post-transplant, cumulative relapse rates at 1 year and 2 years post-transplant, 1-year and 2-year overall survival (OS), graft-versus-host disease-free, relapse-free survival (GRFS), non-relapse mortality (NRM), cumulative incidence of chronic GVHD, and the incidence of Cytomegalovirus （CMV）and Epstein-Barr virus（EBV）reactivation within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and less than 70 years, regardless of gender
* Peripheral T-cell lymphoma (PTCL) was diagnosed according to the 2016 WHO criteria and met any of the following criteria: Relapse: Except ALK+ anaplastic large cell lymphoma （ALCL), CR was achieved by standard chemotherapy but disease progressed，and relapse after hematopoietic stem cell transplantation;Refractory: Except ALK+ anaplastic large cell lymphoma （ALCL), the tumor shrank < 50% or progressive disease after 4 courses of standard chemotherapy, or not achieve CR after 6 courses of standard chemotherapy;Not suitable for or refusing autologous hematopoietic stem cell transplantation.
* Patients must have a suitable hematopoietic stem cell donor:Related donors must have at least 5/10 matches for HLA-A, -B, -C, -DQB1, and - DRB1;Unrelated donors must have at least 8/10 matches for HLA-A, -B, -C, -DQB1, and -DRB1
* Hematopoietic cell transplantation comorbidity index (HCT-CI) score ≤ 2
* ECOG (Eastern Cooperative Oncology Group) performance status: 0-2
* Adequate liver, kidney, and cardiopulmonary function, meeting the following requirements:Serum creatinine ≤ 1.5x ULN (the upper limit of normal);Cardiac function: Ejection fraction ≥ 50%;Baseline oxygen saturation > 92%;Total bilirubin ≤ 2.0 x ULN; ALT and AST ≤ 2.0 x ULN，AKP ≤ 2.0 x ULN;Pulmonary function: DLCO (corrected for hemoglobin) ≥ 40% and FEV1 (Forced Expiratory Volume in 1 second) ≥ 50%
* Patients must have the ability to understand and be willing to participate in this study and sign an informed consent form

Exclusion Criteria:

* PTCL patients did not meet the criteria of relapse / refractory.
* Refuse to adopt allegeneic hematopoietic stem cell transplantation.
* History of malignancies other than lymphoid tumors within the 5 years prior to screening, except for adequately treated in situ cervical cancer, basal cell carcinoma, squamous cell carcinoma of the skin, and curatively treated localized prostate cancer or ductal carcinoma in situ
* ECOG ≥ 3.
* HCT-CI score ≥ 3.
* Any unstable systemic diseases, including but not limited to unstable angina, recent cerebrovascular accidents or transient ischemic attacks within the 3 months prior to screening, myocardial infarction within the 3 months prior to screening, congestive heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias requiring drug treatment after pacemaker implantation, significant liver, kidney, or metabolic diseases, and pulmonary arterial hypertension.
* Active, uncontrolled infections, including those associated with hemodynamic instability, new or worsening infection symptoms or signs, new infectious lesions on imaging, or persistent unexplained fever without signs or symptoms of infection.
* HIV-infected individuals.
* Active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral therapy.
* History of autoimmune diseases
* Pregnant or breastfeeding women.
* Fertile males and females unwilling to use contraception during the treatment period and for 12 months after treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
1y and 2y-progression-free survival (PFS) | up to 1 years for the 1y-PFS and up to 2 years for the 2y-PFS
  1-year and 2-year progression-free survival (PFS) rates post-transplant

SECONDARY OUTCOMES:
acute graft-versus-host disease (aGVHD) | up to 180 days
  acute graft-versus-host disease (aGVHD) within 180 days post-transplant
1y and 2y-cumulative relapse rates (CIR) | up to 1 years for the 1y-CIR and up to 2 years for the 2y-CIR
  cumulative relapse rates (CIR) at 1 year and 2 years post-transplant
1y and 2y-overall survival (OS) | up to 1 years for the 1y-OS and up to 2 years for the 2y-OS
  overall survival (OS) at 1 year and 2 years post-transplant
graft-versus-host disease-free, relapse-free survival (GRFS) | up to 2 years
  graft-versus-host disease-free, relapse-free survival (GRFS) at 2 years post-transplant
non-relapse mortality (NRM) | up to 2 years
  non-relapse mortality (NRM) at 2 years post-transplant
cumulative incidence of chronic GVHD | up to 2 years
  cumulative incidence of chronic GVHD at 2 years post-transplant
CMV and EBV reactivation | up to 1 year
  the incidence of CMV and EBV reactivation within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, MD, Principal Investigator — Shanghai General HospitalShanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao C, Feng J, Gu H, Tang H, Xu L, Dong H, Dong B, Shu M, Bai Q, Liang R, Zhang T, Yang L, Wang Z, Chen X, Gao G. Distribution of lymphoid neoplasms in Northwest China: Analysis of 3244 cases according to WHO classification in a single institution. Ann Diagn Pathol. 2018 Jun;34:60-65. doi: 10.1016/j.anndiagpath.2017.05.005. Epub 2017 May 12. PMID 29661730
- [Background] Yang QP, Zhang WY, Yu JB, Zhao S, Xu H, Wang WY, Bi CF, Zuo Z, Wang XQ, Huang J, Dai L, Liu WP. Subtype distribution of lymphomas in Southwest China: analysis of 6,382 cases using WHO classification in a single institution. Diagn Pathol. 2011 Aug 22;6:77. doi: 10.1186/1746-1596-6-77. PMID 21854649
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] Liu X, Yang M, Wu M, Zheng W, Xie Y, Zhu J, Song Y, Liu W. A retrospective study of the CHOP, CHOPE, and CHOPE/G regimens as the first-line treatment of peripheral T-cell lymphomas. Cancer Chemother Pharmacol. 2019 Mar;83(3):443-449. doi: 10.1007/s00280-018-3744-z. Epub 2018 Dec 3. PMID 30511217
- [Background] Janikova A, Chloupkova R, Campr V, Klener P, Hamouzova J, Belada D, Prochazka V, Pytlik R, Pirnos J, Duras J, Mocikova H, Bortlicek Z, Kopalova N, Mayer J, Trneny M. First-line therapy for T cell lymphomas: a retrospective population-based analysis of 906 T cell lymphoma patients. Ann Hematol. 2019 Aug;98(8):1961-1972. doi: 10.1007/s00277-019-03694-y. Epub 2019 May 8. PMID 31065733
- [Background] Couto SCF, Kowes A, Aurabi CS, Oliveira TGM, Klinger P, Rocha V. Autologous, allogeneic hematopoietic cell transplantation and CAR-T/NK therapy: what is their real importance in PTCL? Front Oncol. 2023 Aug 30;13:1195759. doi: 10.3389/fonc.2023.1195759. eCollection 2023. PMID 37711206
- [Background] Rodriguez J, Caballero MD, Gutierrez A, Marin J, Lahuerta JJ, Sureda A, Carreras E, Leon A, Arranz R, Fernandez de Sevilla A, Zuazu J, Garcia-Larana J, Rifon J, Varela R, Gandarillas M, SanMiguel J, Conde E. High-dose chemotherapy and autologous stem cell transplantation in peripheral T-cell lymphoma: the GEL-TAMO experience. Ann Oncol. 2003 Dec;14(12):1768-75. doi: 10.1093/annonc/mdg459. PMID 14630683
- [Background] Bellei M, Foss FM, Shustov AR, Horwitz SM, Marcheselli L, Kim WS, Cabrera ME, Dlouhy I, Nagler A, Advani RH, Pesce EA, Ko YH, Martinez V, Montoto S, Chiattone C, Moskowitz A, Spina M, Biasoli I, Manni M, Federico M; International T-cell Project Network. The outcome of peripheral T-cell lymphoma patients failing first-line therapy: a report from the prospective, International T-Cell Project. Haematologica. 2018 Jul;103(7):1191-1197. doi: 10.3324/haematol.2017.186577. Epub 2018 Mar 29. PMID 29599200
- [Background] Garcia-Sancho AM, Bellei M, Lopez-Parra M, Gritti G, Cortes M, Novelli S, Panizo C, Petrucci L, Gutierrez A, Dlouhy I, Bastos-Oreiro M, Sancho JM, Ramirez MJ, Moraleda JM, Carrillo E, Jimenez-Ubieto AI, Jarque I, Orsucci L, Garcia-Torres E, Montalban C, Dodero A, Arranz R, De Las Heras N, Pascual MJ, Lopez-Jimenez J, Spina M, Re A, De Villambrosia SG, Bobillo S, Federico M, Caballero D. Autologous stem-cell transplantation as consolidation of first-line chemotherapy in patients with peripheral T-cell lymphoma: a multicenter GELTAMO/FIL study. Haematologica. 2022 Nov 1;107(11):2675-2684. doi: 10.3324/haematol.2021.279426. PMID 35320921
- [Background] Civallero M, Schroers-Martin JG, Horwitz S, Manni M, Stepanishyna Y, Cabrera ME, Vose J, Spina M, Hitz F, Nagler A, Montoto S, Chiattone C, Skrypets T, Perez Saenz MA, Priolo G, Luminari S, Lymboussaki A, Pavlovsky A, Marino D, Liberati M, Trotman J, Mannina D, Federico M, Advani R. Long-term outcome of peripheral T-cell lymphomas: Ten-year follow-up of the International Prospective T-cell Project. Br J Haematol. 2024 Jul;205(1):166-174. doi: 10.1111/bjh.19433. Epub 2024 Mar 26. PMID 38532575
- [Background] Fossard G, Broussais F, Coelho I, Bailly S, Nicolas-Virelizier E, Toussaint E, Lancesseur C, Le Bras F, Willems E, Tchernonog E, Chalopin T, Delarue R, Gressin R, Chauchet A, Gyan E, Cartron G, Bonnet C, Haioun C, Damaj G, Gaulard P, Fornecker L, Ghesquieres H, Tournilhac O, da Silva MG, Bouabdallah R, Salles G, Bachy E. Role of up-front autologous stem-cell transplantation in peripheral T-cell lymphoma for patients in response after induction: an analysis of patients from LYSA centers. Ann Oncol. 2018 Mar 1;29(3):715-723. doi: 10.1093/annonc/mdx787. PMID 29253087
- [Background] Ahn SY, Jung SY, Jung SH, Ahn JS, Lee JJ, Kim HJ, Kang SR, Han YH, Kwak JY, Yhim HY, Yang DH. Prognostic significance of FDG-PET/CT in determining upfront autologous stem cell transplantation for the treatment of peripheral T cell lymphomas. Ann Hematol. 2020 Jan;99(1):83-91. doi: 10.1007/s00277-019-03867-9. Epub 2019 Dec 6. PMID 31807859
- [Background] Schmitz N, Truemper L, Bouabdallah K, Ziepert M, Leclerc M, Cartron G, Jaccard A, Reimer P, Wagner E, Wilhelm M, Sanhes L, Lamy T, de Leval L, Rosenwald A, Roussel M, Kroschinsky F, Lindemann W, Dreger P, Viardot A, Milpied N, Gisselbrecht C, Wulf G, Gyan E, Gaulard P, Bay JO, Glass B, Poeschel V, Damaj G, Sibon D, Delmer A, Bilger K, Banos A, Haenel M, Dreyling M, Metzner B, Keller U, Braulke F, Friedrichs B, Nickelsen M, Altmann B, Tournilhac O. A randomized phase 3 trial of autologous vs allogeneic transplantation as part of first-line therapy in poor-risk peripheral T-NHL. Blood. 2021 May 13;137(19):2646-2656. doi: 10.1182/blood.2020008825. PMID 33512419
- [Background] Loirat M, Chevallier P, Leux C, Moreau A, Bossard C, Guillaume T, Gastinne T, Delaunay J, Blin N, Mahe B, Dubruille V, Augeul-Meunier K, Peterlin P, Maisonneuve H, Moreau P, Juge-Morineau N, Jardel H, Mohty M, Moreau P, Le Gouill S. Upfront allogeneic stem-cell transplantation for patients with nonlocalized untreated peripheral T-cell lymphoma: an intention-to-treat analysis from a single center. Ann Oncol. 2015 Feb;26(2):386-92. doi: 10.1093/annonc/mdu515. Epub 2014 Nov 12. PMID 25392158
- [Background] Rohlfing S, Dietrich S, Witzens-Harig M, Hegenbart U, Schonland S, Luft T, Ho AD, Dreger P. The impact of stem cell transplantation on the natural course of peripheral T-cell lymphoma: a real-world experience. Ann Hematol. 2018 Jul;97(7):1241-1250. doi: 10.1007/s00277-018-3288-7. Epub 2018 Mar 16. PMID 29549411